CLINICAL TRIAL: NCT03351049
Title: An RCT on Support Surfaces for Pressure Ulcer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Brienza (Other)
Responsible Party: Sponsor-Investigator, David Brienza, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO16030036
Record Dates: First submitted 2017-11-15; First posted 2017-11-22 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Pressure Injury; Pressure Ulcer
Keywords: Acute care, support surface
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Reactive, Low air loss support surface (Experimental): Participants in this arm will use a reactive support surface with a low air loss feature
  Interventions: Device: LAL
- Reactive, non-low air loss (Active Comparator): Participants in this arm will use a reactive support surface without a low air loss feature
  Interventions: Device: Non-LAL

INTERVENTIONS:
Device: LAL — Reactive support surface with a low air loss feature
  Arms: Reactive, Low air loss support surface
Device: Non-LAL — Reactive support surface without a low air loss feature
  Arms: Reactive, non-low air loss

SUMMARY:
Pressure injuries are a serious health care problem and affect millions of people. Most pressure injuries are avoidable with the application of best practices and with the use of appropriate technology. Support surfaces are a crucial component of any comprehensive prevention strategy. Decades of research have produced moderate and low levels of evidence upon which to base clinical decisions concerning how and when to apply support surfaces for prevention. This knowledge has been periodically assessed and assembled into clinical practice guidelines. There is good evidence that the combined group of active and reactive support surfaces is effective in preventing pressure injuries and that high-specification reactive foam surfaces are effective in preventing pressure injuries. But there is insufficient evidence that low air loss surfaces are more or less effective than other types of surfaces. Yet, low air loss surfaces are used for more than 17% of patients in acute care at high risk of developing pressure injuries.

The study is designed to determine if and when low air loss is effective in preventing pressure injuries, and what level of heat and moisture control performance is necessary for prevention effectiveness. The primary aim of the project is to compare the effectiveness of reactive support surfaces with low air loss to reactive support surfaces without low air loss in preventing pressure injuries for people with moisture risk factors in acute care. Support surfaces are currently marketed and identified by practitioners based on device features (e.g., low air loss, air fluidization, alternating pressure), categories (powered, non-powered, reactive, and active) and components (e.g., foam, gel, fluid).

The critical performance characteristics of low air loss systems are moisture, humidity and temperature management. Preliminary work has revealed that these characteristics vary widely among different low air loss products. A secondary aim of the proposed study is to explore associations between support surface performance characteristics and pressure injury outcomes to identify which low air loss performance characteristics and what level of those performance characteristics are necessary for the technology to be effective.

Successful completion of this project will fill a critical gap in evidence regarding the effectiveness of support surfaces with low air loss, and could influence a shift in the way support surfaces are characterized away from the current feature-based paradigm toward a more clinically relevant and generalizable performance-based paradigm.

DETAILED DESCRIPTION:
Pressure injuries are a serious health care problem and threaten the health and well-being of millions of people. Most pressure injuries are avoidable with the application of standard practices and proper utilization of existing technology. Support surface technology has been shown to prevent pressure injuries, but the effectiveness of specific features designed for management of tissue loads, microclimate (i.e., heat and moisture), and/or other therapeutic functions are unknown. Preclinical research has demonstrated that heat and moisture are important pressure injury risk factors. Low air loss is a support surface feature designed to manage the heat and moisture at the interface between the person and the surface. It is a feature that is invariably combined with the provision of pressure redistribution through immersion and envelopment. Clinical research has produced evidence to support the use of reactive support surfaces with good immersion and envelopment characteristics, but there is a gap in evidence regarding the effectiveness of microclimate management features.

This study aims to first determine if low air loss is effective for preventing pressure injuries. Second, to facilitate translation of the results to clinical practice, the study is designed to identify which low air loss performance characteristics and what levels of those performance characteristics are necessary for the technology to be effective.

Aim 1 will compare the effectiveness of reactive support surfaces with low air loss to reactive support surfaces without low air loss in preventing pressure injuries for people with moisture risk factors in acute care. This aim will also investigate the comparative effectiveness in subgroups defined by age, body mass index (BMI), Braden score, and Braden mobility subscale score. We will also investigate the association between pressure injury severity and treatment group.

Aim 2 will explore associations between support surface performance characteristics and pressure injury outcomes. Performance will be quantified by the microclimate control measures of evaporative capacity and heat flux.

An individual randomized design with 816 subjects will be used to achieve the aims. Participants will be randomized into either a low air loss or no-low air loss surface type across seven possible groups differentiated only by the support surface assignment. The seven surfaces will have a range of heat and moisture control performance characteristics. Biological variables, pressure injury incidence, pressure injury risk factors and related clinical conditions and procedures will be recorded and analyzed. For Aim 2, to explore associations between support surface performance characteristics and pressure injuries, we will determine threshold and cutoff values for optimum effectiveness.

The proposed study is designed to fill a critical gap in evidence regarding the effectiveness of support surfaces with low air loss. The study will also explore cutoff scores or ranges of effective performance for microclimate control. If successful, the study could influence a shift in the way support surfaces are characterized away from the current feature-based paradigm toward a more accurate and generalizable performance-based paradigm.

Study protocol: An individual randomized design will be used to achieve the aims. The study procedures and flow is depicted in Figure 1. Eligible acute care patients will be identified and enrolled within 24 hours of admission. New admissions will be screened for the following criteria for inclusion: 1. total Braden score≤18 and 2. Braden Moisture sub-scale score 1-constantly moist or 2-very moist, 3. projected length of stay ≥4 days, and 4. absence of pressure injuries.

After informed consent, absence of pressure injuries will be confirmed, baseline data (demographic and clinical data) will be recorded and participants will be randomized to one of seven groups differentiated only by the support surface assignment. The seven surfaces can be divided into reactive support surface with low air loss (5 total) or reactive surface without low air loss (2 total) for analyses of Aim 1, and demonstrate a range of heat and water vapor control performance characteristics for analyses of Aim 2. Once enrolled, the participant will be provided the intervention within 24 hours.

Participants in all groups will be provided usual care including tissue integrity management according to UPMC system-wide Skin Integrity Procedures, which address risk assessment (daily), skin inspection (twice daily), regular patient repositioning (every two hours as condition allows), pressure alleviation, moisture control, nutritional support and friction/shear relief applications. Outcomes will be recorded from electronic medical records and through assessment by research staff until pressure injury incidence or hospital discharge.

The outcome measures were chosen to ensure direct relevance to patients at risk for developing pressure injuries. We chose the direct clinical outcome measure of pressure injury incidence to assess the clinical effectiveness of the study support surface interventions being compared.

Pressure injury status will be assessed daily. Pressure injury risk factors, ambulatory status and related preventive interventions (support surface related conditions such as layers of linens, and interventions such as turning schedules) will be monitored and recorded every day (7 days per week) from electronic medical records, observation by research staff and interviews with clinical staff until any of the following endpoints are reached: pressure injury incidence, Braden score >18, or discharge from hospital. After an endpoint is reached, length of stay, and, for participants that develop pressure injuries, the severity will be recorded as the highest injury stage reached prior to discharge (Stage 1, 2, 3, 4, DTPI or unstageable) as defined by the National Pressure Ulcer Advisory Panel. If the injury status was observed to be a DTPI or unstageable at any point in time and later becomes identified as 1, 2, 3, or 4, the latter stage will be recorded. Otherwise DTPIs and unstageable injuries will be recorded as such.

Variables believed to be associated with the study outcome of pressure injuries include: 1. Demographic and clinical characteristics: age, race, ethnicity, weight, height, and medical comorbidities such as diabetes, peripheral vascular disease, nutritional status, and incontinence. These will be recorded at baseline. 2. Pressure injury risk factors: Braden score, Braden sub-scale scores, and ambulatory status will be monitored and recorded daily until endpoint. 3. Clinical conditions and procedures: layers of linens, interventions such as turning schedules, and type and length of the surgery will be monitored and recorded daily until endpoint. 4. Length of stay and number of days on the support surface will be recorded at study endpoint.

816 participants will be identified and recruited from the adult inpatient population of facilities in the University of Pittsburgh hospital system (UPMC).

The study will use a 2:1 allocation randomization scheme stratifying by support surface type (2 LAL to 1 no-LAL). The rationale for having a 2:1 allocation is to allow us to achieve both aims. The 2:1 allocation is necessary because we plan to randomize to 5 LAL groups and 2 no-LAL groups. We will use randomized blocks of varying length (containing random permutations of the two surface types, LAL vs. no LAL, across the seven groups) for randomization. T.

ELIGIBILITY:
Inclusion Criteria:

* total Braden Score <= 18
* Braden Moisture sub-scale score 1 or 2
* projected length of stay in hospital >= 4 days
* absent of pressure injuries

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Brienza, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian and Montefiore, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based upon chart review at 1 academic medical center between September 2018 and April 2022.
Pre-assignment Details: Of 457 enrolled participants, 451 met inclusion criteria and were randomized.
Period: Overall Study
Arm/Group | Reactive, Low Air Loss Support Surface | Reactive, Non-low Air Loss
Started | 323 | 128
Completed | 297 | 106
Not Completed | 26 | 22
Not completed — Withdrawal | 26 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reactive, Low Air Loss Support Surface | Reactive, Non-low Air Loss | Total
Number analyzed (Participants) | 323 | 128 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (13.8) | 68.3 (14.5) | 67.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 73 | 230
  Male | 166 | 55 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 247 | 96 | 343
  Unknown or Not Reported | 74 | 32 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 240 | 95 | 335
  Black | 46 | 24 | 70
  Other | 7 | 0 | 7
  Missing | 30 | 9 | 39
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28 (7) | 29 (7) | 28 (7)
Braden Score [Mean (Standard Deviation); unit: units on a scale] — Pressure injury/ulcer risk assessment tool. The scale consists of six subscales and the total scores range from 6-23. The six subscales include sensory, moisture, activity, mobility, nutrition, friction/shear. A lower Braden score indicates higher levels of risk for pressure injury development.
  units on a scale | 13.8 (2.2) | 13.8 (2.2) | 13.8 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Pressure Injury
Description: Number of participants who had a new pressure injury occur during study participation
Time Frame: Through study completion, an average of 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reactive, Low Air Loss Support Surface | Reactive, Non-low Air Loss
Number analyzed (Participants) | 323 | 128
Participants | 23 | 10
Statistical Analysis 1: Comparison: Reactive, Low Air Loss Support Surface vs Reactive, Non-low Air Loss; Compare the effectiveness of reactive support surfaces with and without low air loss in preventing pressure injuries; Test type: Superiority; p = 0.8, Chi-squared

ADVERSE EVENTS:
Time Frame: Over entire period of study intervention which varied due to variations in number of days in the hospital. The average number of days for the treatment group was 11 and for the control group was 10.
Arm/Group | Reactive, Low Air Loss Support Surface | Reactive, Non-low Air Loss
All-Cause Mortality (participants affected / at risk) | 0/323 | 0/128
Serious Adverse Events (participants affected / at risk) | 0/323 | 0/128
Other Adverse Events (participants affected / at risk) | 0/323 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03351049/Prot_SAP_001.pdf